CLINICAL TRIAL: NCT02520752
Title: A Phase I, Multicenter, Open-label, Single-sequence Drug-drug Interaction Study to Assess the Effect of INC280 on the Pharmacokinetics of Midazolam and Caffeine in Patients With cMET-dysregulated Advanced Solid Tumors
Brief Title: A DDI Study to Assess the Effect of INC280 on the PK of Midazolam and Caffeine in Patients With cMET-dysregulated Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2103
Record Dates: First submitted 2015-08-09; First posted 2015-08-13 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-07

CONDITIONS: cMET-dysregulated Advanced Solid Tumors
Keywords: cMET, INC280, caffeine, midazolam
MeSH Terms: interventions — capmatinib; Midazolam; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INC280 (Experimental)
  Interventions: Drug: INC280; Drug: Midazolam; Drug: Caffeine

INTERVENTIONS:
Drug: INC280
Drug: Midazolam
Drug: Caffeine

SUMMARY:
Drg-drug Interaction (DDI) study to assess the effect of INC280 on the pharmacokinetics of midazolam and caffeine in patients with cMET-dysregulated advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

Patients must have:

* advanced solid tumors and have confirmed cMET dysregulation
* at least one measurable lesion as defined by RECIST 1.1.
* recovered from all toxicities related to prior anti-cancer therapies
* adequate organ function
* ECOG performance status (PS) of 0 or 1

Exclusion Criteria:

Patients must not have:

* known hypersensitivity to any of the excipients of INC280 or to benzodiazepines or known intolerance and hypersensitivity to caffeine
* symptomatic central nervous system (CNS) metastases who are neurologically unstable
* presence or history of carcinomatous meningitis
* history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Clinically significant, uncontrolled heart diseases, including QTcF ≥ 450 ms (male patients), ≥ 460 ms (female patients) on the screening ECG
* Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting INC280
* Major surgery within 4 weeks prior to starting INC280
* Patients receiving unstable or increasing doses of corticosteroids.
* Impairment of GI function or GI disease that may significantly alter the absorption of INC280
* Patients who have received or consumed, or are expected to receive or consume midazolam or caffeine-containing products (e.g., tea, coffee, cola), within 2 days prior to Day 1 and during the whole duration of the DDI phase (i.e., from Day -2 to Day 12)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
AUClast of midazolam and caffeine | Up to 72 hours post midazolam and caffeine dose
  midazolam and caffeine pharmacokinetic parameters
AUCinf of midazolam and caffeine | Up to 72 hours post midazolam and caffeine dose
  midazolam and caffeine pharmacokinetic parameter
Lambda_z of midazolam and caffeine | Up to 72 hours post midazolam and caffeine dose
  midazolam and caffeine pharmacokinetic parameter
Cmax of midazolam and caffeine | Up to 72 hours post midazolam and caffeine dose
  midazolam and caffeine pharmacokinetic parameter
Tmax of midazolam and caffeine | Up to 72 hours post midazolam and caffeine dose
  midazolam and caffeine pharmacokinetic parameter
T1/2 of midazolam and caffeine | Up to 72 hours post midazolam and caffeine dose
  midazolam and caffeine pharmacokinetic parameter
CL/F of midazolam and caffeine | Up to 72 hours post midazolam and caffeine dose
  midazolam and caffeine pharmacokinetic parameter
Vz/F of midazolam and caffeine | Up to 72 hours post midazolam and caffeine dose
  midazolam and caffeine pharmacokinetic parameter

SECONDARY OUTCOMES:
Adverse events based on the CTCAE v4.03 grade (severity) and other safety data (e.g.,ECG, vital signs, laboratory results) | From consent to 30 days post last dose
  To assess safety and tolerability of INC280 in patients with cMET-dysregulated advanced solid tumors
Overall response rate of patients treated with INC280 | Baseline, every 6 weeks
  Overall response rate is defined as Complete Response and Partial Response calculated per RECIST 1.1, per investigator assessment
Disease control rate of patients treated with INC280 | Baseline, every 6 weeks
  Disease control rate is defined as calculated as the proportion of patients with best overall response of Complete Response, Partial Response, or Stable Disease calculated per RECIST 1.1, per investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (2):
  - Emory University School of Medicine/Winship Cancer Institute SC-2, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Copenhagen, Denmark
- France (2):
  - Novartis Investigative Site, Dijon, Cote D Or
  - Novartis Investigative Site, Pierre-Bénite
- Novartis Investigative Site, Rozzano, MI, Italy
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CINC280A2103 can be found on the Novartis Clinical trial results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17184